CLINICAL TRIAL: NCT05324111
Title: VaLidation of the Simple Adaptation of the Kardia 6L ECG Recorder to Obtain Chest leAd equivaLents: a Multi-centre International (LOCAL-ECG) Study; on Behalf of the Africa Heart Rhythm Association Investigators
Acronym: LOCAL-ECG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CD21/140756
Record Dates: First submitted 2022-03-31; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 12 Lead ECG (Experimental): Application of hand held electrocardio gram
  Interventions: Device: Kardia 6L

INTERVENTIONS:
Device: Kardia 6L — The Kardia 6L has CE marking. The purpose of this study is to extend the use of this device by a simple modification using existing equipment in the department. The device will be connected to the left leg electrodes using standard clinical crocodile clips and the other electrode applied to the chest in V1 and V6 positions to acquire the modified V1 and V6 leads

SUMMARY:
ECGs are routinely performed in cardiology. Recently handheld ECGs have shown promise in screening for heart rhythm disorders. These are quick to perform and do not require the preparation that is needed for 12 lead ECGs. The aim is to test whether a novel adaptation to a handheld ECG recorder, Kardia 6L, which has the potential to record a 6 lead ECG is able to screen for ECG abnormalities, thereby obviating the need for a full 12 lead ECG. This may allow for earlier diagnosis and treatment and has implications in the prevention of infection.

The lead author recently published a pilot study showing the clinical utility of this technique and the aim of this study is to validate the method.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who is attending the cardiology clinic or an inpatient on the cardiology ward who consents to taking part

Exclusion Criteria:

* Patients who are unable or refuse to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-08-04 (Actual); Primary Completion 2023-02-07 (Estimated); Study Completion 2023-02-07 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of adaptation to handheld 6Lead | 10 Minutes
  Sensitivity and specificity of adaptation to handheld 6Lead compared to 12 lead for leads V1 and V6 for the measurement of PR, QRS duration and QT interval

SECONDARY OUTCOMES:
Assessment of other ECG parameters | 10 Minutes
  Assessment of other ECG parameters e.g. ST segment change in the ECG wave

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospital NHS Trust, Leeds, United Kingdom